CLINICAL TRIAL: NCT03210545
Title: A Dose-response Study of Markers of Glucocorticoid Effects (DOSCORT): A Double-blinded, Randomized, 2-dose, Cross-over Study
Brief Title: A Study of Markers of Glucocorticoid Effects in Patients With Addisons Disease (DOSCORT)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DOSCORT; 2016-004078-16 (EudraCT Number)
Record Dates: First submitted 2017-06-29; First posted 2017-07-07 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Addison Disease
Keywords: Biomarker; Glucocorticoids; Metabolism
MeSH Terms: conditions — Addison Disease | interventions — Betamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- betamethasone - physiological dose (Active Comparator): Replacing participants hydrocortisone with a daily dose of betamethasone in an estimated physiological dose during one treatment period.
  Interventions: Drug: Betamethasone
- betamethasone - supra physiological dose (Active Comparator): Replacing participants hydrocortisone with a daily dose of betamethasone in an estimated supra physiological dose during one treatment period.
  Interventions: Drug: Betamethasone

INTERVENTIONS:
Drug: Betamethasone — A cross-over study where patients with Addison´s disease will undergo two treatment periods where their usual hydrocortisone replacement therapy will be replaced by the glucocorticoid betamethasone in physiological and supra physiological doses. A wash-out period of 2-5 weeks in-between the treatment periods will be carried out where participants intake their usual hydrocortisone replacement therapy.

SUMMARY:
DOSCORT is a 2-dose, cross-over study primarily aiming to identify and validate novel biological markers (biomarkers) of glucocorticoid effect in the human body. Patients with Addison´s disease, primary adrenal insufficiency, with life-long glucocorticoid replacement therapy will undergo 2 treatment periods where their usual hydrocortisone treatment will be replaced with betamethasone in physiological and supra physiological doses. Blood, saliva, urine, health related Quality-of-life self-assessment forms, measurements of physical activity and sleep quality will be collected from both treatment periods.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females at ages 20-65 years
2. Previously diagnosed (e.g. more than 12 months ago) with primary adrenal insufficiency due to autoimmune adrenalitis, i.e. Addison´s disease
3. A stable daily glucocorticoid replacement dose for at least 3 months prior to study entry
4. An oral glucocorticoid replacement dose of 15-30 mg Hydrocortisone total daily dose
5. If needed, a stable fludrocortisone replacement dose for at least 3 months prior to study entry
6. Body mass index (BMI) of 20-35 kg/m2
7. Ability to comply to the protocol procedures and having signed informed consent to participate in the study

Exclusion Criteria:

1. Clinical or laboratory signs of significant cerebral, cardiovascular, respiratory, hepaticobiliary/ pancreatic disease which in the investigators judgement may interfere with the study assessment of completion of the study
2. Clinically significant renal dysfunction with a serum creatinine above 150 mmol/L
3. Pregnant or lactating women
4. Diabetes Mellitus
5. Systemic infections
6. Regular dehydroepiandrosterone (DHEA) medication for the past 4 weeks
7. Any medication with agents which in the investigators judgement might interfere with the study drugs kinetics, including therapies affecting gastro intestinal emptying or motility
8. Alcohol/drug abuse or any other condition associated with poor patient compliance, including expected non-cooperation, as judged by the investigator
9. Hypersensitivity to the active substance or any excipients used in the study drug of choice
10. Any additional underlying disease that may need regular or periodic pharmacological treatment with glucocorticoids during the trail, such as asthma, skin- or eye conditions treated with inhaled or topical glucocorticoids
11. Any additional underlying condition that needs treatment with intramuscular or intra-articular steroid injections during the trial

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Protein profile changes between physiological and supra physiological doses of betamethasone. | Changes in proteome (g/dl or umol/l) during 7 days of treatment with two different doses of betamethasone
  By using mas spectrometry, protein profile changes in blood, urine and saliva will be identified at four timepoints: after 3 hours and after 7 days during treatment with betamethasone in a physiological dose and after 3 hours and after 7 days during treatment with betamethasone in a supra physiological dose.
Metabolite profile changes between physiological and supra physiological doses of betamethasone. | Changes in metabolome (units depending on the kind of metabolome) during 7 days of treatment with two different doses of betamethasone
  By using mas spectrometry, metabolite profile changes in blood, urine and saliva will be identified at four timepoints: after 3 hours and after 7 days during treatment with betamethasone in a physiological dose and after 3 hours and after 7 days during treatment with betamethasone in a supra physiological dose.

SECONDARY OUTCOMES:
Messenger RNA (mRNA)/miRNA profile changes between physiological and supra physiological doses of betamethasone. | Changes in mRNA/miRNA (Svedberg Unit, S) during 7 days of treatment with two different doses of betamethasone
  By using array based transcriptomics (both mRNA and miRNA), mRNA/miRNA profile changes in blood, urine and saliva will be identified at four timepoints: after 3 hours and after 7 days during treatment with betamethasone in a physiological dose and after 3 hours and after 7 days during treatment with betamethasone in a supra physiological dose.
Changes in glucose metabolism between physiological and supra physiological doses of betamethasone. | Changes in glucose metabolism (units depending on sample analysis) during 7 days of treatment with two different doses of betamethasone
  Conventional markers for glucose metabolism in blood will be identified at four timepoints: after 3 hours and after 7 days during treatment with betamethasone in a physiological dose and after 3 hours and after 7 days during treatment with betamethasone in a supra physiological dose.
Changes in lipid-profile between physiological and supra physiological doses of betamethasone. | Changes in lipid-profile (units depending on sample analysis) during 7 days of treatment with two different doses of betamethasone
  Conventional markers for lipid-profile in blood will be identified at four timepoints: after 3 hours and after 7 days during treatment with betamethasone in a physiological dose and after 3 hours and after 7 days during treatment with betamethasone in a supra physiological dose.
Changes in bone-markers between physiological and supra physiological doses of betamethasone. | Changes in levels of bone-markers in blood (units depending on sample analysis) during 7 days of treatment with two different doses of betamethasone
  Bone-markers in blood will be identified at four timepoints: after 3 hours and after 7 days during treatment with betamethasone in a physiological dose and after 3 hours and after 7 days during treatment with betamethasone in a supra physiological dose.
Changes in self-reported Quality of Life between physiological and supra physiological doses of betamethasone using the Addison-specific Quality of Life questionnaire (ADDIQoL). | Changes in units of the ADDIQoL questionnaire (units on a scale) after 7 days of treatment with two different doses of betamethasone
  Self-reported health-related quality of life and general well-being will be assessed using the ADDIQoL questionnaire after 7 days of treatment with a physiological dose of betamethasone and after 7 days of treatment with a supra physiological dose of betamethasone.
Changes in self-reported Quality of Life between physiological and supra physiological doses of betamethasone using the Psychological General Well-being (PGWB) index. | Changes in units of the PGWB index (units on a scale) after 7 days of treatment with two different doses of dexamethasone
  Self-reported health-related quality of life and general well-being will be assessed using the PGWB index after 7 days of treatment with a physiological dose of betamethasone and after 7 days of treatment with a supra physiological dose of betamethasone.
Changes in self-reported quality of life and fatigue between physiological and supra physiological doses of betamethasone using the Fatigue impact scale (FIS) | Changes in units in the FIS (units on a scale) after 7 days of treatment with two different doses of betamethasone
  Self-reported health-related quality of Life, general well-being and fatigue will be assessed using the FIS questionnaire after 7 days of treatment with a physiological dose of betamethasone and after 7 days of treatment with a supra physiological dose of betamethasone.
Changes in self-reported quality of life and fatigue between physiological and supra physiological doses of betamethasone using the Functional Outcomes of Sleep Questionnaire (FOSQ). | Changes in units in the FOSQ (units on a scale) after 7 days of treatment with two different doses of betamethasone
  Self-reported health-related quality of life, general well-being and fatigue will be assessed using FOSQ after 7 days of treatment with a physiological dose of betamethasone and after 7 days of treatment with a supra physiological dose of betamethasone.
Changes in daily physical activity between physiological and supra physiological doses of betamethasone | Changes in daily physical activity (units provided in connected software) after 7 days of treatment with two different doses of betamethasone
  Daily physical activity will be objectively evaluated using a wrist accelerometer during 7 days of treatment with a physiological dose of betamethasone and during 7 days of treatment with a supra physiological dose of betamethasone.
Changes in sleep quality between physiological and supra physiological doses of betamethasone | Changes in sleep quality (measurements and units provided in connected software) after 7 days of treatment with two different doses of betamethasone
  Sleep quality will be objectively evaluated using a wrist worn sleep monitor during the last night of a 7 day treatment period with a physiological dose of betamethasone and the last night of a 7 day treatment period with a supra physiological dose of betamethasone.

CONTACTS AND LOCATIONS:
Overall Officials: Gudmundur Johannsson, Prof., MD, Principal Investigator — Vastra Gotaland Region, Sahlgrenska University Hospital, dept. of Endocrinology
Locations (1):
- Centrum for Endocrinology and Metabolism, Sahlgenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided